CLINICAL TRIAL: NCT00394927
Title: A Multicenter, Non-interventional Surveillance Study to Evaluate the Adverse Effects of Antiepileptic Drug Treatment in Patients With Epilepsy
Brief Title: Adverse Event Scale in Patients With Epilepsy (aEscape) - A European Survey for Physicians With Epilepsy Patients
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Collaborators: International Bureau for Epilepsy (Other)
Other Study IDs: N01228
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Epilepsy
Keywords: Non-Interventional; Surveillance; Adverse Effects; AntiEpileptic Drug treatment
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort

SUMMARY:
The purpose of the survey is to explore through a structured interview and patient examination the rate and distribution of neurological and systemic adverse effects related to antiepileptic treatment. Adverse effects and considerations to modify the therapy will be assessed in pediatric and adult patients with controlled as well as uncontrolled epilepsy with different seizure types

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients from the age of 4 years
* Confirmed diagnosis of epilepsy requiring AED treatment
* Patients already receiving daily AED treatment as a monotherapy or a polytherapy with maximum 2 AEDs within the terms of marketing authorization with the following medications: Carbamazepine, Clobazam, Clonazepam, Gabapentin, Lamotrigine, Levetiracetam, Oxcarbazepine, Phenobarbital, Phenytoin, Pregabalin, Tiagabine, Topiramate, Valproate, Zonisamide
* Treatment must be stable for at least 3 months prior to assessment
* Absence of other severe and/or uncontrolled symptomatic chronic illness

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed diagnosis of epilepsy requiring anti-epileptic treatment and which are already receiving daily anti-epileptic treatment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Buyle, M.D., Study Director — UCB Pharma
Locations (53):
- Vienna, Austria
- Czechia (15):
  - Blansko
  - České Budějovice
  - Hradec Králové
  - Karlovy Vary
  - Kopřivnice
  - Kroměříž
  - Liberec
  - Litomyšl
  - Náchod
  - Nové Město na Moravě
  - Prague
  - Teplice
  - Třebíč
  - Ústí nad Labem
  - Zlín
- Germany (16):
  - Aschaffenburg
  - Berlin
  - Bielefeld
  - Bochum
  - Cologne
  - Düsseldorf
  - Ellwangen
  - Göttingen
  - Hirschaid
  - Jena
  - Königsbrück
  - Krefeld
  - Leipzig
  - München
  - Neuberg
  - Oelde
- Italy (2):
  - Albano Laziale (Roma)
  - Napoli
- Poland (10):
  - Bialystok
  - Elblag
  - Gdansk
  - Katowice
  - Kielce
  - Krakow
  - Lublin
  - Poznan
  - Warsaw
  - Wroclaw
- Romania (8):
  - Botoșani
  - Brasov
  - Bucharest
  - Craiova
  - Galati
  - Iași
  - Lasi
  - Timișoara
- Sant Boi de Llobregat, Spain